CLINICAL TRIAL: NCT02287012
Title: Quantification of the Time and Effort Required for Peripheral Blood Stem Cell Collection - The European Perspective
Brief Title: Quantification of the Time and Effort Required for Peripheral Blood Stem Cell Collection -The European Perspective
Status: Completed | Type: Observational
Sponsor: Pr Mohamad MOHTY (Other)
Responsible Party: Sponsor-Investigator, Pr Mohamad MOHTY, Professor, Association for Training, Education, and Research in Hematology, Immunology, and Transplantation
Organization: Association for Training, Education, and Research in Hematology, Immunology, and Transplantation (Other)
Other Study IDs: Mozo Time and Motion
Record Dates: First submitted 2014-11-03; First posted 2014-11-10 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-01

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pre-Plerixafor era: The first era (Pre-Plerixafor era) will be defined as a two year period immediately preceding commercialization of plerixafor in Europe, (e.g., June 1, 2007 through June 1, 2009).
- Plerixafor era: The second era (Plerixafor era) will be defined as July 1, 2010 through July 1, 2012).
  Interventions: Other: Time/Motion evaluation of actual apheresis

INTERVENTIONS:
Other: Time/Motion evaluation of actual apheresis — The actual apheresis events will be measured in consecutive patients scheduled to be candidates for peripheral blood stem mobilization in the apheresis area of the hospital. Each apheresis will be considered as one event . Should the patient receive more than 1 apheresis, each apheresis will be considered as one different event.
  Groups: Plerixafor era

SUMMARY:
This study aims to observe the effects of the availability of plerixafor on the time and effort associated with autologous peripheral blood stem cell collection.

DETAILED DESCRIPTION:
This non interventional study will consist of two parts:

I. Retrospective study:

A medical record review will be conducted covering 200 patients file undergoing peripheral blood stem cell mobilization in some European centers.

II. Prospective study :Time/Motion evaluation of actual apheresis - 20 events each center The actual apheresis events will be measured in consecutive patients scheduled to be candidates for peripheral blood stem mobilization in the apheresis area of the hospital. Each apheresis will be considered as one event . Should the patient receive more than 1 apheresis, each apheresis will be considered as one different event.

ELIGIBILITY:
Inclusion Criteria:

Patients must satisfy the following for the part 1

* Oncology patients diagnosed with Non-Hodgkin lymphoma who are candidates for autologous hematopoietic stem cell transplantation (HSCT)
* A patient that fails to achieve a target CD34+>20 cells/µl, before or on the first day of apheresis
* Age > 18 years

Exclusion Criteria for the part 1

Patients with:

* Age < 18 years;
* Primary diagnosis other than Non-Hodgkin lymphoma
* Undergone prior autologous hematopoietic stem cell transplantation (HSCT)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will consist of two parts:
  I. Retrospective study:
  A medical record review will be conducted covering 200 patients file undergoing peripheral blood stem cell mobilization in different European centers. Patients will be selected from each of centers, evenly divided between two eras: 1) prior to approval of plerixafor= Pre-P era (July 2009); and 2) after approval of plerixafor= P era .
  II. Prospective study :Time/Motion evaluation of actual apheresis - 20 events each center
Sampling Method: Non-Probability Sample
Enrollment: 248 (Actual)
Dates: Start 2013-10; Primary Completion 2015-06 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Type, duration and length of administration of mobilizing agents | one week
  Number of visits for administration of mobilizing agents Duration (days) of administration of mobilizing agents Type of agents used as mobilizing agents
Number and length of apheresis sessions and number of collected stem cells | one week
  Number of apheresis sessions Number of hours of apheresis sessions Attainment of CD34+ cells target (yes, no) Number of days until CD34+ target level is met

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad Mohty, MD, PhD, Principal Investigator — Hôpital Saint-Antoine